CLINICAL TRIAL: NCT04998929
Title: A Common But Unknown Disease; A Case Series Study
Brief Title: A Common But Unknown Disease; Nave Sliding (NS)
Acronym: NS
Status: Completed | Type: Observational
Sponsor: Komar University of Science and Technology (Other)
Responsible Party: Principal Investigator, yosra raziani, principal investigator,nursing department, lecturer, Komar University of Science and Technology
Other Study IDs: Komar
Record Dates: First submitted 2021-07-28; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-07

CONDITIONS: Navel; Hernia
Keywords: nave sliding; abdominal wall defect
MeSH Terms: conditions — Hernia | interventions — Complementary Therapies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: complementary therapy — traditional techniques of treatment including, (a)cupping therapy, (b)Backstroke for young people, (c)Sitting on all fours while the other person holds both knees firmly with the hands, the patient is asked to bend at the back so that the abdominal muscles are stretched, (d)taking a nerve that passes under the armpit with two index fingers and thumbs and applying intense pressure to the extent that the patient goes unconscious due to the severity of the pain, (e)Hanging the patient from the horizontal bar and stretching the abdominal muscles, (f)Tie an onion-sized object such as, a bag of wheat or salt, with a scarf on the navel for one hour, (g) taking the gum of mountain pistachio tree which is the same as turpentine and halve a walnut and fill it with raw turpentine and put it inside the navel for 72 hours, and then move it in the umbilical region by twisting hand movements, (h)cupping therapy.

SUMMARY:
The present study is a case series study, conducted to introduce a common disease of abdominal wall which has received less attention in scientific resources. The study population was all patients who following repeated hospital visits did not improve, and for their last try, they visited a traditional clinic, and were diagnosed with umbilical hernia.

DETAILED DESCRIPTION:
Background: The present study is conducted to introduce a common disease of abdominal wall which has received less attention in scientific resources. In traditional medicine sources Some scholars believe that this condition occurs due to the movement of the abdominal muscle near the umbilicus or nave laterally movement of nave.

Design: A case series study Method: This study was a case series study. The study population was all patients who following repeated hospital visits did not improve, and for their last try, they visited a traditional clinic, and were diagnosed with umbilical hernia during a period of 5 months.

ELIGIBILITY:
inclusion Criteria:

* Clinical diagnosis of nave sliding
* Must be able to provide a complete health history information

Exclusion Criteria:

* unwillingness to continue
* any unexpected complication of traditional treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 20 patients who following repeated hospital visits did not improve, and for their last try, they visited a traditional clinic, and were diagnosed with nave sliding
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Demographic information questionnaire | 1 hour through study completion
  age, gender
standard form of health history taking | 5 hour through study completion
  onset of the disease, cause, signs and symptoms, Hospital visits and all medical procedures, including lab test results, imaging, failed medical interventions that the patients have received once they suspected the problem with their health, and differential diagnosis.
body mass index | once at admission time
  BMI in kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Komar University, Sulaymaniyah, Iran, Iraq

IPD SHARING:
Plan to Share IPD: No